CLINICAL TRIAL: NCT06279689
Title: Measurement of Skin-to-Muscle and Skin-to-Bone Distances in Adult and Pediatric Populations Before and While Applying a Force Similar to the ZENEO® Triggering Force
Brief Title: Echography Study_Anthropometric Measurements
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Crossject (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CJTCDZ2301
Record Dates: First submitted 2024-01-31; First posted 2024-02-28 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects : Adult and pediatric populations (Experimental): Only ultrasound procedures will be performed using an investigational ultrasound system.
  All subjects will be asked to undergo 1 on site visit (Study Visit) during which the eligibility assessment and the ultrasound scans will be performed is to evaluate the anatomical characteristics of both anterolateral thighs, one shoulder (deltoid) and one upper arm (biceps and triceps) before and while applying a force similar to the ZENEO® triggering force.
  Interventions: Other: Ultrasound scans

INTERVENTIONS:
Other: Ultrasound scans — Ultrasound scans connected with an application enabling the measurement of the force applied.

SUMMARY:
This is a multi-center, exploratory, estimation study in both adult and pediatric populations. There is no investigational product injection during this study The exploratory objective of this study is to evaluate the anatomical characteristics of both anterolateral thighs in healthy adult and healthy pediatric populations (2 to 17 years old) by ultrasound scan before and while applying a force similar to the ZENEO® triggering force.

In the healthy adult population, anatomical characteristics of one shoulder (deltoid) and one upper arm (biceps and triceps) will also be evaluated by ultrasound scan before and while applying a force similar to ZENEO® triggering force.

Only ultrasound procedures will be performed using an investigational ultrasound system. All subjects will be asked to undergo 1 on site visit (Study Visit) during which the eligibility assessment and the ultrasound scans will be performed.

DETAILED DESCRIPTION:
The exploratory endpoints are as follows:

* The skin-to-muscle distance (STMD) (mm) before and while applying a force on both anterolateral thighs, one shoulder (deltoid), and one upper arm (biceps and triceps) in the adult population and both anterolateral thighs in the pediatric population
* The skin-to-bone distance (STBD) (mm) before and while applying a force on both anterolateral thighs, one shoulder (deltoid), and one upper arm (biceps and triceps) in the adult population and both anterolateral thighs in the pediatric population
* The thickness of skin layers (mm) (thickness of dermis, thickness of hypodermis [ie, subcutaneous fat]) before and while applying a force on both anterolateral thighs, one shoulder (deltoid), and one upper arm (biceps and triceps) in the adult population and both anterolateral thighs in the pediatric population
* The thickness of muscle layers (mm) before and while applying a force on both anterolateral thighs, one shoulder (deltoid), and one upper arm (biceps and triceps) in the adult population and both anterolateral thighs in the pediatric population

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 2 to 70 years old, inclusive
2. In stable health, as determined by medical history and physical examination at screening (ie, any chronic medical diagnoses or conditions should be stable and well managed, with no significant changes expected during assessments, so that in the opinion of the investigator or designee there will not be any impact on the ability of the subject to participate in the study)
3. For the adult population, body mass index (BMI) ≥ 18.5 and ≤ 35 kg/m2 at screening BMI = weight (kg)/(height [m])2
4. Willing and able to provide written informed consent and assent (as appropriate) prior to initiation of study procedures
5. Subjects must be able to communicate effectively with the study staff and to understand study instructions (not applicable for toddlers and preschoolers)

Exclusion Criteria:

1. Any skin or muscular condition, such as eczema, scars, infections, moles, or tattoos at the site of measurements
2. Allergy to ultrasound gel
3. Any other condition or prior therapy that, in the investigator or designee's opinion, would make the subject unsuitable for the study, or unable or unwilling to comply with the study procedures
4. Is an employee or authorized representative of CROSSJECT SA or ICON plc
5. Adult under guardianship or subject incarcerated

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
STBD : Skin To Bone Distance | Day1
  Distance measurement
STMD: Skin To Muscle Distance | Day1
  Distance measurement
Thickness of skin layers (dermis, hypodermis) | Day1
  Thickness measurement
Thickness of muscle layers | Day1
  Thickness measurement

SECONDARY OUTCOMES:
Circumferences measurements (thigh, upper arm, waist, hip) | Day1
  Measurement

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie LOUGHRAIEB, Study Director — Crossject
Locations (1):
- Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No